CLINICAL TRIAL: NCT00719706
Title: The Use of a Mitochondrial Enhancement Treatment in Bipolar Disorder: A Randomized, Placebo-Controlled Trial of Acetyl-L-Carnitine and Alpha-Lipoic Acid for the Treatment of Bipolar Depression
Brief Title: The Use of a Mitochondrial Enhancement Treatment in Bipolar Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Brian P. Brennan, MD, Associate Director of Translational Neuroscience Research, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008-P-000772
Record Dates: First submitted 2008-07-18; First posted 2008-07-22 (Estimated); Results first posted 2012-07-18 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-06

CONDITIONS: Bipolar Depression
Keywords: Bipolar disorder; Bipolar depression; Natural substances; Depression
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — Acetylcarnitine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 1000-3000mg/day of acetyl-l-carnitine PLUS 600-1800mg/day of alpha-lipoic acid
  Interventions: Drug: acetyl-l-carnitine PLUS alpha-lipoic acide
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: acetyl-l-carnitine PLUS alpha-lipoic acide — 1000-3000 mg/day of acetyl-l-carnitine in addition to 600-1800 mg/day of alpha-lipoic acid.
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
The primary objective of this 15-week clinical trial is to test the hypothesis that treatment with two proven mitochondrial enhancers, acetyl-L-carnitine (ALCAR) and α-lipoic acid (ALA), has significantly greater efficacy than placebo as an augmentation treatment in bipolar depressed patients who display an incomplete response to conventional treatments.

DETAILED DESCRIPTION:
The primary objective of this proposed clinical trial is to test the hypothesis that treatment with two proven mitochondrial enhancers, acetyl-L-carnitine (ALCAR) and α-lipoic acid (ALA), has significantly greater efficacy than placebo as an augmentation treatment in bipolar depressed patients who display an incomplete response to conventional treatments. We propose to test this hypothesis by performing a 15-week placebo-controlled, double-blind, parallel group, flexible-dose study investigating the use of ALCAR and ALA as an augmentation to treatment as usual in depressed bipolar patients. We will compare the efficacy of acetyl-l-carnitine (ALCAR) at doses of 1000-3000mg/day and alpha-lipoic acid (ALA) at doses of 600-1800mg/day with placebo on symptom improvement in individuals diagnosed with bipolar disorder type I, current episode depressed. Improvement will be assessed using the 21-Item Hamilton Depression Rating Scale (HAM-D), the Montgomery Asberg Depression Rating Scale (MADRS), the Young Mania Rating Scale (YMRS), and the Clinical Global Impression-Severity and Improvement Scales (CGI-S and CGI-I).

Furthermore, we hypothesize that improvement in depression symptoms following treatment with ALCAR and ALA will be associated with increases in phosphocreatine (PCr), beta-nucleoside triphosphate (β-NTP), and intracellular pH in the anterior cingulate cortex (ACC) both at week 1 and week 12 of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18-65 years.
* Meets DSM-IV criteria for Bipolar Disorder, type I with current episode depressed.
* Current score of greater than or equal to 18 on the 21-Item Hamilton Depression Rating Scale at Visits 1 and 2.
* Maintained on a stable treatment regimen with no changes in medication dosages for at least two weeks prior to study entry.

Exclusion Criteria:

* Unwilling or unable to provide informed consent
* Score of greater than or equal to 12 on the Young Mania Rating Scale at Visit 1 or 2.
* Current suicidal or homicidal ideation.
* Active psychotic symptoms.
* Lifetime history of schizophrenia or obsessive-compulsive disorder.
* DSM-IV diagnosis of alcohol or substance dependence in the 3 months prior to screening.
* Clinically significant medical condition that would interfere with study participation.
* History of hypersensitivity to ACLCAR or ALA.
* Pregnant or lactating.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-08; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian P Brennan, MD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in August 2008 and ended in May 2011 and took place at a research lab within McLean hospital.
Pre-assignment Details: To limit heterogeneity in the imaging sample, we accepted only type I bipolar disorder participants for the imaging component of the study.
Groups:
- ALCAR/ALA: Participants taking 1000-3000mg/day of acetyl-l-carnitine PLUS 600-1800mg/day of alpha-lipoic acid.
- Placebo: Participants taking placebo.
Period: Overall Study
Arm/Group | ALCAR/ALA | Placebo
Started | 20 | 20
Completed | 11 | 14
Not Completed | 9 | 6
Not completed — Adverse Event | 5 | 4
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Protocol Violation | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ALCAR/ALA | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 46 (10.3) | 44.9 (11.9) | 45.45 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 9 | 7 | 16
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: The 25-Item Hamilton Depression Rating Scale.
Description: Scores could range from 0 - 72 units on a scale, with 0 representing the least number of depressive symptoms and 72 representing the most number of depressive symptoms.
Time Frame: Baseline to 15 Weeks
Population: At baseline, the number of participants analyzed was the number randomized into the study. At endpoint, the number or participants analyzed is the last observation carried forward of the original 20 participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ALCAR/ALA | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale
  Baseline Data | 23.3 (3.5) | 22.1 (3.2)
  Endpoint Data | 17.5 (6.4) | 18.5 (6.2)

2. Primary Outcome: The Montgomery-Asberg Depression Rating Scale
Description: Scores could range from 0 - 60 units on a scale with 0 representing the least number of depressive symptoms and 60 representing the most number of depressive symptoms.
Time Frame: Baseline to 15 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ALCAR/ALA | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale
  Baseline Data | 26.9 (3.1) | 25.9 (3)
  Endpoint Data | 19.6 (7.9) | 21.7 (6.3)

3. Primary Outcome: The Young Mania Rating Scale
Description: The scores could range from 0 - 60 units on a scale with 0 representing the least number of manic symptoms and 60 representing the most number of manic symptoms.
Time Frame: Baseline to 15 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ALCAR/ALA | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale
  Baseline Data | 2 (2.1) | 2.4 (2.1)
  Endpoint Data | 1.7 (2.2) | 2.1 (1.8)

4. Primary Outcome: Clinical Global Impression-Severity
Description: Scores could range from 0 - 7 units on a scale, with 0 representing the least severe ("Normal, not at all ill") and 7 representing the most severe ("Among the most extremely ill patients").
Time Frame: Baseline to 15 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ALCAR/ALA | Placebo
Number analyzed (Participants) | 20 | 20
units on a scale
  Baseline Data | 4.6 (0.5) | 4.6 (0.51)
  Endpoint Data | 4 (0.9) | 4.2 (0.7)

5. Secondary Outcome: Phosphorus MRS Scans on 4T Scanner
Description: Whole brain total NTP levels as measured by a phosphorus MRS scan on the 4T scanner. The data could range from 0 - 1, with 0 representing the lowest NTP level and 1 representing the highest NTP level.
Time Frame: Baseline to 12 weeks
Population: At baseline, the number of participants analyzed was the number entered into the imaging portion of the study. At endpoint, the number or participants analyzed is the last observation carried forward of the original 10 participants in each category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ALCAR/ALA | Placebo
Number analyzed (Participants) | 10 | 10
units on a scale
  Baseline Data | .230 (.009) | .233 (.009)
  Week 1 Data | .229 (.011) | .225 (.008)
  Endpoint Data | .229 (.006) | .232 (.005)

ADVERSE EVENTS:
Time Frame: Baseline to 13 weeks.
Arm/Group | ALCAR/ALA | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 20/20 | 19/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ALCAR/ALA (N=20) | Placebo (N=20)
diarrhea (Gastrointestinal disorders) | 6 | 3
foul-smelling urine (Renal and urinary disorders) | 5 | 1
rash (Skin and subcutaneous tissue disorders) | 4 | 0
constipation (Gastrointestinal disorders) | 3 | 1
dyspepsia (Gastrointestinal disorders) | 3 | 0
nausea (Gastrointestinal disorders) | 2 | 5
abdominal cramping (Gastrointestinal disorders) | 2 | 3
chest pain (Cardiac disorders) | 2 | 0
restlessness (General disorders) | 2 | 1
pruritis (Skin and subcutaneous tissue disorders) | 2 | 1
vomiting (Gastrointestinal disorders) | 2 | 0
sedation (General disorders) | 2 | 0
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 | 2
dry mouth (General disorders) | 2 | 1
insomnia (General disorders) | 1 | 5
flu-like illness (Gastrointestinal disorders) | 1 | 0
fatigue (General disorders) | 1 | 0
headache (General disorders) | 1 | 3
blood in stool (Gastrointestinal disorders) | 1 | 0
blurred vision (Eye disorders) | 1 | 0
word-finding difficulties (Psychiatric disorders) | 1 | 0
hirsuitism (Endocrine disorders) | 1 | 0
facial flushing (Vascular disorders) | 1 | 0
decreased taste (General disorders) | 1 | 0
salty taste (General disorders) | 1 | 0
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
dizziness (General disorders) | 1 | 1
flatulence (Gastrointestinal disorders) | 0 | 4
anxiety (Psychiatric disorders) | 0 | 1
sore throat (General disorders) | 0 | 1
facial acne (Skin and subcutaneous tissue disorders) | 0 | 1
irritability (Psychiatric disorders) | 0 | 2
bloating (Gastrointestinal disorders) | 0 | 1
weight gain (General disorders) | 0 | 2
tremor (General disorders) | 0 | 1
urinary frequency (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes